CLINICAL TRIAL: NCT05434598
Title: A Prospective Study of Whole Genome Sequencing (ChromoSeq) as an Adjunct to Conventional Genomic Profiling in MDS
Brief Title: Whole Genome Sequencing (ChromoSeq) as an Adjunct to Conventional Genomic Profiling in MDS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: American Society of Hematology (Other); Edward P. Evans Foundation (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 202206077; UH3CA272904 (NIH)
Record Dates: First submitted 2022-06-21; First posted 2022-06-28 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Whole Genome Sequencing; Myelodysplastic Syndromes
MeSH Terms: conditions — Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Patients: ChromSeq (Experimental): ChromoSeq will be performed on bone marrow or peripheral blood DNA from consented patients in parallel with the standard of care cytogenetics, FISH, and the MyeloSeq gene panel obtained from that sample, in a CLIA licensed environment using CLIA-compliant ChromoSeq procedures.
  Interventions: Device: ChromoSeq
- Stakeholders (Treating Physicians) (No Intervention): Stakeholders (treating physicians) will complete surveys/questionnaires

INTERVENTIONS:
Device: ChromoSeq — Novel, streamlined whole genome sequencing approach
  Arms: Patients: ChromSeq

SUMMARY:
This is a single institution, prospective study of the whole genome sequencing assay, ChromoSeq. Using prospectively collected patient data, coupled with physician surveys, the investigators seek to determine the feasibility of implementing ChromoSeq in addition to standard genomic testing, for patients with the diagnosis of myelodysplastic syndrome (MDS).

ELIGIBILITY:
Inclusion Criteria Patient:

* Diagnosis of MDS, or a clinical suspicion for a new diagnosis of MDS, for whom routine diagnostic testing is requested or planned to be requested.
* Seen in the outpatient setting.
* Not been previously treated with disease-modifying therapy (such as lenalidomide or hypomethylating agents).

Note: Patients who have received transfusional support, erythropoietin-stimulating agents, growth factor support, or luspatercept are eligible.

At least 18 years of age.

-Able to understand and willing to sign an IRB approved written informed consent document.

Inclusion Criteria Physician:

* Treating physician at Washington University School of Medicine who directs therapy for individuals with hematologic malignancies.
* Able and willing to complete standardized questionnaires about stakeholder perceptions of ChromoSeq during the ChromoSeq implementation process. (Written documentation of informed consent is not required.)

Exclusion Criteria Patient:

-Younger than 18 years of age

Exclusion Criteria Physician

-Does not treat patients at Washington University School of Medicine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-27 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Rate of assay success on first attempt between ChromoSeq and conventional cytogenetics as measured by total number of recurrent structural variants identified | Through completion of all ChromoSeq tests (estimated to be 24 months)
  -The number of recurrent structural variants detected by ChromoSeq will be compared to those detected by conventional cytogenetics using two non-inferiority tests for dependent samples using non-inferiority margin of 1%.
Rate of assay success on first attempt between ChromoSeq and conventional cytogenetics as measured by total number of copy number alterations identified | Through completion of all ChromoSeq tests (estimated to be 24 months)
  The number of copy number alterations detected by ChromoSeq will be compared to those detected by conventional cytogenetics using two non-inferiority tests for dependent samples using non-inferiority margin of 1%.
Proportion of failed ChromoSeq assays | Through completion of all ChromoSeq tests (estimated to be 24 months)
  * As compared to failed standard of care genomic profiling assays
  * The proportion of first-run failures for ChromoSeq assays will be compared to the proportion of failed standard of care genomic profiling assays using a directional Fisher's exact test.

SECONDARY OUTCOMES:
Stakeholder perceptions of ChromoSeq | Through 1 month after generation of ChromoSeq for all patients enrolled (estimated to be 25 months)
  * Using survey responses from treating physicians obtained from per case standardized questionnaires designed using Consolidated Framework for Implementation Research constructs
  * For each case, the corresponding treating physician will be asked to answer a case-based ChromoSeq Implementation Physician Survey. In order to prospectively investigate how the ChromoSeq data was used or could be used by the treating physician for each case, and to evaluate perceptions in real time, the physician will be asked to complete the survey within 1 month of the ChromoSeq and completed conventional genomic profiling results being returned to the chart, whichever is later.

CONTACTS AND LOCATIONS:
Overall Officials: Meagan A Jacoby, M.D., Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 3 months and ending 5 years following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal may submit proposals to mjacoby@wustl.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu